CLINICAL TRIAL: NCT01873495
Title: Omacetaxine for Consolidation and Maintenance in Patients Age ≥ 55 With AML in First Remission: A Pilot Study
Brief Title: Omacetaxine for Consolidation and Maintenance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Martha Arellano, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057844; Winship2176-11 (Other: Other)
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acute Myelogenous Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omacetaxine: Consolidation/Maintenance (Experimental)
  Interventions: Drug: Omacetaxine

INTERVENTIONS:
Drug: Omacetaxine — Omacetaxine 1.25 mg/m² sub-cutaneously twice daily for 5 consecutive days every 28 (± 8) days for 3 cycles.
  Patients in continuous remission after 3 cycles of consolidation will receive maintenance omacetaxine 1.25 mg/m² twice daily for 3 days, every 28 days for up to 6 cycles
  Other Names: Synribo

SUMMARY:
The purpose of this pilot study is to assess the safety and tolerability of omacetaxine for consolidation in patients age 55 and older with acute myelogenous leukemia (AML) in first complete remission following induction with cytarabine and an anthracycline, and also to assess the safety and tolerability of omacetaxine for maintenance in patients age 55 and older with acute AML in first complete remission following 3 consolidation courses with omacetaxine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML including de novo, secondary, or with an antecedent hematologic disorder (AHD) according to the World Health Organization (WHO) criteria.
2. Age ≥ 55 years.
3. Patient eligible for standard induction chemotherapy based on Eastern Cooperative Oncology Group (ECOG) performance status and vital organ function at the discretion of the treating physician.
4. Patients who received 1-2 cycles of hypomethylating therapy (decitabine azacitidine) are eligible.
5. Provide signed written informed consent.
6. Be able to comply with study procedures and follow-up examinations.
7. Be non-fertile or agree to use birth control during the study through the end of last treatment visit.
8. Adequate renal and hepatic function at the time of second registration:

   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); and
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; and
   * Serum creatinine ≤ 1.2 x ULN.
9. ECOG performance ≤ 2 at the time of second registration.
10. Patients with a history of carcinoma in remission, on no therapy or on hormonal therapy for the adjuvant treatment of breast carcinoma or prostate carcinoma are included in the study.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL, French-American-British [FAB] classification M3 or WHO classification of APL with t (15;17)(q22;q12), (PML/retinoic acid receptor alpha [RARa] and variants).
2. Prior treatment with omacetaxine.
3. Relapsed or refractory AML.
4. Investigational agent received within 30 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 2 or less prior to first dose of study drug.
5. Psychiatric disorders that would interfere with consent, study participation, or follow-up.
6. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
7. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo the proposed therapy. This includes uncontrolled hypertension and uncontrolled diabetes, as cases of life threatening hyperglycemia have been reported (using continuous infusion at higher doses of omacetaxine).
8. Active carcinoma requiring systemic chemotherapy or radiation therapy.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha L. Arellano, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 5/8/2013 and 7/23/2018 at Winship Cancer Institute of Emory University.
Period: Overall Study
Arm/Group | Omacetaxine: Consolidation/Maintenance
Started | 7
Completed | 0
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1
Not completed — Removed for Transplantation | 1
Not completed — AML (Acute Myelogenous Leukemia) Relapse | 1

BASELINE CHARACTERISTICS:
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease Status Assessment Prior to Each Consolidation Cycle
Description: Disease status will be assessed by a bone marrow aspirate and biopsy prior to each of 3 consolidation cycles (to ensure that patients are still in remission).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 7
Participants
  Relapsed AML | 0
  Remission | 7

2. Primary Outcome: Assessment of Disease Status
Description: Bone marrow biopsy and aspirate will be obtained.
Time Frame: 1 month
Population: Seven patients completed at least one cycle of omacetaxine.
Measure: Count of Participants; unit: Participants
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 7
Participants
  Relapsed AML | 1
  Remission | 6

3. Primary Outcome: Bone Marrow Aspirate to Confirm Continuous Remission
Description: Bone marrow aspirate to confirm continuous remission will be obtained before starting maintenance and at 3 and 6 months from the start of maintenance.
Time Frame: 3 months
Population: No patients entered the maintenance phase of this study.
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 0

4. Primary Outcome: Maintenance Toxicities
Description: Toxicities will be monitored by history, physical examination, and laboratory monitoring during maintenance.
Time Frame: 24 weeks
Population: No patients entered the maintenance phase of this study.
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 0

5. Secondary Outcome: Consolidation Toxicities
Description: Toxicities will be monitored by history, physical examination, and laboratory monitoring (CBC, serum chemistries to include renal and liver function tests) obtained weekly during consolidation and monthly during maintenance according to standard of care (Appendices C and D). Toxicity will be assessed according to the NCI Common Toxicity Criteria Version 4.0 (available at the NCI web site http://ctep.cancer.gov/reporting/ctc.html).
Time Frame: 12 weeks
Population: Two participants experienced toxicities: thrombocytopenia and atrial flutter.
Measure: Count of Participants; unit: Participants
Arm/Group | Omacetaxine: Consolidation/Maintenance
Number analyzed (Participants) | 7
Participants
  Thrombocytopenia | 1
  Atrial Flutter | 1
  No Toxicities | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly during consolidation and monthly during maintenance.
Arm/Group | Omacetaxine: Consolidation/Maintenance
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omacetaxine: Consolidation/Maintenance (N=7)
Atrial flutter (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omacetaxine: Consolidation/Maintenance (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Accrual was halted early due to the inability of 30% of subjects to complete the intended consolidation and maintenance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT01873495/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT01873495/ICF_001.pdf